CLINICAL TRIAL: NCT01138111
Title: ß-amyloid Imaging With BAY94-9172 Positron Emission Tomography for Early Detection of Alzheimer's Disease in Patients With Mild Cognitive Impairment
Brief Title: Florbetaben (BAY94-9172) PET (Positron Emission Tomography) Imaging in MCI (Mild Cognitive Impairment) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 312043
Record Dates: First submitted 2010-04-01; First posted 2010-06-07 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-05

CONDITIONS: Alzheimer Disease; Amyloid Beta-Protein
Keywords: Florbetaben; Amyloid beta-protein; MCI; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Florbetaben (BAY94-9172)

INTERVENTIONS:
Drug: Florbetaben (BAY94-9172) — single 300 megabecquerel (MBq) intravenous injection 2 mL to 10 mL, at baseline, at 12 and 24 months

SUMMARY:
The aim of the study is to investigate whether Florbetaben (BAY94-9172)positron emission tomography (PET) is able to distinguish between subjects with mild cognitive impairment (MCI) progressing to Alzheimer's disease (AD) from those with MCI not progressing to AD.

ELIGIBILITY:
Inclusion Criteria:

* Presence of MCI defined as abnormal cognition on objective testing in the absence of dementia or significant functional loss.
* Absence of systemic or other neurological disease that may contribute to cognitive impairment or prevent follow-up over two years.
* Able to give written informed consent.
* Age >/= 60 years of age
* >/= 7 years of education

Exclusion Criteria:

* Mini mental state examination (MMSE) score < 24 at baseline
* Clinical dementia rating (CDR) score > 0.5 at baseline
* Patients who receive regular medication of drugs which may adversely impact cognition (e.g. tricyclic antidepressants, antipsychotics and/or large doses of hypnotics or anxiolytics)
* Existing or history of cancer
* History of severe head trauma, brain surgery or intracranial hematoma with permanent brain lesion
* Lifetime history of major affective disorder, schizophrenia, or schizo-affective disorder
* Contraindications to MRI (Magnetic resonance imaging)
* Relevant history, physical or imaging findings of neurological disease other than MCI and mild depression
* History of severe anaphylactic reaction or high risk of allergic reaction to drugs
* Patient has received another investigational drug in the preceding 14 days

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Heidelberg, Victoria, Australia

REFERENCES:
- [Derived] Bullich S, Roe-Vellve N, Marquie M, Landau SM, Barthel H, Villemagne VL, Sanabria A, Tartari JP, Sotolongo-Grau O, Dore V, Koglin N, Muller A, Perrotin A, Jovalekic A, De Santi S, Tarraga L, Stephens AW, Rowe CC, Sabri O, Seibyl JP, Boada M. Early detection of amyloid load using 18F-florbetaben PET. Alzheimers Res Ther. 2021 Mar 27;13(1):67. doi: 10.1186/s13195-021-00807-6. PMID 33773598
- [Derived] Ong KT, Villemagne VL, Bahar-Fuchs A, Lamb F, Langdon N, Catafau AM, Stephens AW, Seibyl J, Dinkelborg LM, Reininger CB, Putz B, Rohde B, Masters CL, Rowe CC. Abeta imaging with 18F-florbetaben in prodromal Alzheimer's disease: a prospective outcome study. J Neurol Neurosurg Psychiatry. 2015 Apr;86(4):431-6. doi: 10.1136/jnnp-2014-308094. Epub 2014 Jun 26. PMID 24970906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 71 patients were screened at one study center in Australia. The first subject's consent was obtained on 02 JUN 2008.
Pre-assignment Details: 26 subjects were screen failures and did not have study drug administered.
Groups:
- MCI Subjects: Subjects with mild cognitive impairment (MCI) receiving florbetaben (BAY94-9172) : single intravenous injection of 300 megaBecqerels (MBq) florbetaben, at baseline, at 12 and 24 months
Period: Overall Study
Arm/Group | MCI Subjects
Started | 45
Completed | 36
Not Completed | 9
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who received at least one florbetaben (BAY94-9172) injection
Groups:
- MCI Subjects: Subjects with mild cognitive impairment (MCI) receiving florbetaben (BAY94-9172) : single intravenous injection 2 mL to 10 mL, at baseline, at 12 and 24 months
Arm/Group | MCI Subjects
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 29
Region of Enrollment [Number; unit: participants]
  Australia | 45

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Assessment of Neocortical SUVRs (Mean Standard Uptake Value Ratios) as a Measure of Florbetaben Uptake
Description: Mean SUVRs were calculated for subjects who did and did not progress to Alzheimer's Disease (AD) during the study for each PET scan time point (baseline, 12 and 24 months)
Time Frame: 1 scanning period post injection to be evaluated at baseline, 12 months and 24 months
Population: All subjects receiving study drug with PET scan data at the respective timepoint
Measure: Mean (Standard Deviation); unit: SUVR
Groups:
- Not Progressed to AD (Baseline): Mean SUVR for the baseline PET scan in subjects who did not progress to AD during the study
- Progressed to AD (Baseline): Mean SUVR for the baseline PET scan in subjects who progressed to AD during the study
- Not Progressed to AD (12 Month): Mean SUVR for the 12 month PET scan in subjects who did not progress to AD during the study
- Progressed to AD (12 Month): Mean SUVR for the 12 month PET scan in subjects who progressed to AD during the study
- Not Progressed to AD (24 Month): Mean SUVR for the 24 month PET scan in subjects who did not progress to AD during the study
- Progressed to AD (24 Month): Mean SUVR for the 24 month PET scan in subjects who progressed to AD during the study
Arm/Group | Not Progressed to AD (Baseline) | Progressed to AD (Baseline) | Not Progressed to AD (12 Month) | Progressed to AD (12 Month) | Not Progressed to AD (24 Month) | Progressed to AD (24 Month)
Number analyzed (Participants) | 26 | 19 | 24 | 17 | 22 | 14
SUVR | 1.430 (0.252) | 1.726 (0.227) | 1.442 (0.270) | 1.738 (0.236) | 1.439 (0.219) | 1.796 (0.296)
Statistical Analysis 1: Comparison: Not Progressed to AD (Baseline) vs Progressed to AD (Baseline); The baseline neocortical SUVR in those subjects who progressed to AD over the 2 year follow-up was compared to the neocortical SUVR of those that did not progress by a Wilcoxon-Mann-Whitney test; Test type: Superiority or Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Not Progressed to AD (12 Month) vs Progressed to AD (12 Month); The 12 month neocortical SUVR in those subjects who progressed to AD over the 2 year follow-up was compared to the neocortical SUVR of those that did not progress by a Wilcoxon-Mann-Whitney test; Test type: Superiority or Other; p = 0.0011, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Not Progressed to AD (24 Month) vs Progressed to AD (24 Month); The 24 month neocortical SUVR in those subjects who progressed to AD over the 2 year follow-up was compared to the neocortical SUVR of those that did not progress by a Wilcoxon-Mann-Whitney test; Test type: Superiority or Other; p = 0.0008, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Normal and Abnormal Scans in Patients With MCI Progressing to AD and Those Who do Not Progress Based on a Threshold of Neocortical SUVR=1.4
Description: This outcome measure showed the number of abnormal scans in subjects with MCI progressing to AD and those who did not progress compared to subjects with normal scans that did not progress and those who did progress.
Time Frame: 1 scanning period post injection to be evaluated at baseline, at 12 months and at 24 months
Population: All subjects receiving study drug
Measure: Number; unit: participants
Groups:
- Not Progressed to AD (Baseline): Results from baseline scan for participants with no progression to AD within 2 years after baseline scan
- Progressed to AD (Baseline): Results from baseline scan for participants with progression from MCI to AD within 2 years after baseline scan.
- Not Progressed to AD (12 Month): Results from 12 month scan for participants with no progression to AD within 2 years after baseline scan.
- Progressed to AD (12 Month): Results from 12 month scan for participants with progression from MCI to AD within 2 years after baseline scan.
- Not Progressed to AD (24 Month): Results from 24 month scan for participants with no progression to AD within 2 years after baseline scan.
- Progressed to AD (24 Month): Results from 24 month scan for participants with progression from MCI to AD within 2 years after baseline scan.
Arm/Group | Not Progressed to AD (Baseline) | Progressed to AD (Baseline) | Not Progressed to AD (12 Month) | Progressed to AD (12 Month) | Not Progressed to AD (24 Month) | Progressed to AD (24 Month)
Number analyzed (Participants) | 26 | 19 | 24 | 18 | 22 | 14
participants
  Number with Normal Scan | 17 | 2 | 15 | 2 | 12 | 1
  Number with Abnormal Scan | 9 | 17 | 9 | 16 | 10 | 13

3. Secondary Outcome: Number and Proportion of Normal and Abnormal Scans Based on Brain ß-amyloid Plaque Load (BAPL) in Subjects With MCI Converting to AD and Those Who do Not Progress
Description: At each study time point (baseline, 12 months and 24 months) PET images were obtained at 45 min and again at 90 post injection. These images were assigned a BAPL score of 1, 2 or 3 based on the reader's evaluation of the scan. A BAPL scores of 1 was considered normal, and scores of 2 and 3 were considered abnormal. These scores were compared to subjects clinical diagnosis for AD at the end of the study follow up period.
Time Frame: 2 scanning periods post injection to be evaluated each at baseline, at 12 months, and at 24 months
Population: All subjects with PET data at the referenced study time point
Measure: Number; unit: participants
Groups:
- Not Progressed to AD (Baseline): Baseline PET scan results for subjects who did not progress to AD through the end of the two year follow up period
- Progressed to AD (Baseline): Baseline PET scan results for subjects who progressed to AD within the two year follow up period
- Not Progressed to AD (12 Month): 12 month PET scan results for subjects who did not progress to AD through the end of the two year follow up period
- Progressed to AD (12 Month): 12 month PET scan results for subjects who progressed to AD within the two year follow up period
- Not Progressed to AD (24 Month): 24 month scan results for subjects who did not progress to AD through the end of the two year follow up period
- Progressed to AD (24 Month): 24 month PET scan results for subjects who progressed to AD within the two year follow up period
Arm/Group | Not Progressed to AD (Baseline) | Progressed to AD (Baseline) | Not Progressed to AD (12 Month) | Progressed to AD (12 Month) | Not Progressed to AD (24 Month) | Progressed to AD (24 Month)
Number analyzed (Participants) | 26 | 19 | 24 | 17 | 22 | 14
participants
  45 min normal PET assessment | 15 | 2 | 16 | 0 | 14 | 0
  45 min abnormal PET assessment | 11 | 17 | 8 | 17 | 8 | 14
  90 min normal PET assessment | 16 | 0 | 14 | 1 | 14 | 2
  90 min abnormal PET assessment | 10 | 19 | 10 | 16 | 8 | 12

4. Secondary Outcome: Sensitivity/Specificity/Negative Predictive Value (NPV)/Positive Predictive Value (PPV) at Baseline, 12, and 24 Months in the Detection of Significant Brain ß-amyloid Plaque Load in Patients With MCI Progressing to AD Compared to Those Who do Not Progress
Description: Sensitivity, specificity, NPV and PPV were measured based on subject BAPL scores by time point and imaging window, compared to clinical diagnosis of AD during the study period. A BAPL score of 1 was considered negative for the presence of beta-amyloid, and scores of 2 and 3 were considered positive.
  For this study, sensitivity was defined as the percentage of subjects with a clinical diagnosis of AD who also had a positive PET scan (BAPL score of 2 or 3) at the respective time point.
  Specificity was defined as the percentage of subjects with a clinical diagnosis of non-AD who also had a negative PET scan (BAPL score of 0 or 1) at the respective time point.
  PPV was defined as the probability that a subject with a positive PET scan would have a clinical diagnosis of AD sometime during the 2 year follow up period.
  NPV was defined as the probability that a subject with a negative PET scan would not have a clinical diagnosis of AD at any point during the 2 year follow up period.
Time Frame: 2 scanning periods post injection to be evaluated at baseline
Population: All subjects with PET data at the referenced study time point
Measure: Number; unit: percentage of subjects
Groups:
- Baseline 45 Min: Baseline PET scan at 45 min post-injection
- Baseline 90 Min: Baseline PET scan at 90 min post-injection
- 12 Month 45 Min: 12 month PET scan at 45 min post-injection
- 12 Month 90 Min: 12 month PET scan at 90 min post-injection
- 24 Month 45 Min: 24 month PET scan at 45 min post-injection
- 24 Month 90 Min: 24 month PET scan at 90 min post-injection
Arm/Group | Baseline 45 Min | Baseline 90 Min | 12 Month 45 Min | 12 Month 90 Min | 24 Month 45 Min | 24 Month 90 Min
Number analyzed (Participants) | 45 | 45 | 41 | 41 | 36 | 36
percentage of subjects
  Sensitivity | 89.47 | 100.00 | 100.00 | 94.12 | 100.00 | 85.71
  Specificity | 57.69 | 61.54 | 66.67 | 58.33 | 63.64 | 63.64
  Positive Predictive value | 60.71 | 65.52 | 68.00 | 61.54 | 63.64 | 60.00
  Negative predictive value | 88.24 | 100.00 | 100.00 | 93.33 | 100.00 | 87.50

ADVERSE EVENTS:
Time Frame: AEs were defined for the period starting immediately after injection and up to the 7 day follow-up (baseline, 12 month, and 24 month follow-up visit.)
Groups:
- MCI Subjects (Initial Drug Administration): Subjects with AEs following the initial administration of florbetaben (BAY94-9172) at the baseline visit
- MCI Subjects (1st Repeat Drug Administration): Subjects with AEs following the second administration of florbetaben (BAY94-9172) at the 12 month visit
- MCI Subjects (2nd Repeat Drug Administration): Subjects with AEs following the third administration of florbetaben (BAY94-9172) at the 24 month visit
Arm/Group | MCI Subjects (Initial Drug Administration) | MCI Subjects (1st Repeat Drug Administration) | MCI Subjects (2nd Repeat Drug Administration)
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/41 | 2/36
Other Adverse Events (participants affected / at risk) | 13/45 | 3/41 | 2/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCI Subjects (Initial Drug Administration) (N=45) | MCI Subjects (1st Repeat Drug Administration) (N=41) | MCI Subjects (2nd Repeat Drug Administration) (N=36)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MCI Subjects (Initial Drug Administration) (N=45) | MCI Subjects (1st Repeat Drug Administration) (N=41) | MCI Subjects (2nd Repeat Drug Administration) (N=36)
Catheter site haemorrhage (General disorders) | 3 (3) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 9 (9) | 0 (0) | 2 (2)
Burning sensation (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less